CLINICAL TRIAL: NCT02780050
Title: Influence of Core Muscles Activation Using Physical Fitness on the Performance of Chest Compression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Choi Hyun Young, Clinical Assistant professor, Hallym University Kangnam Sacred Heart Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-03-26
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Last update posted 2016-06-13 (Estimated); Status verified 2016-06

CONDITIONS: Heart Arrest
Keywords: cardiopulmonary resuscitation; manikins; physical fitness
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chest compression before physical fitness (No Intervention): The subjects consist of 25 medical school students and interns had experienced in cardiopulmonary resuscitation (CPR) education.
  2 instructors, they had physical therapy (PT) certificate, take an exam for subject's muscle strength of each muscle. After that time, subjects take a rest for 10 minutes. Researchers educate to subjects for high quality CPR including 5 to 6cm compression depth, 100 to 120 beat per minute (bpm) rate, complete chest recoil. Subjects perform chest compression to manikin with skill reporting system during 4min under guidance of 110 bpm metronome sound (first chest compression). Researchers record subject's chest compression depth and rate in 1st chest compression.
- after core muscle activation using physical fitness (Experimental): The subjects consist of 25 medical school students and interns had experienced in cardiopulmonary resuscitation (CPR) education.
  After 1st chest compression, subjects take a rest during an hour and carry out PT. PT consist of 30 second plank for 3 sets, 12 times bridge for 3 sets and 20 times leg extension for 3 sets. Subjects take a rest during 30 seconds between sets, 1 minute every 3 sets.
  After PT completion, subjects take a rest during 10 minutes, and then perform 2nd chest compression in the same way of 1st chest compression. Researchers record subject's chest compression depth and rate in 2nd chest compression.
  Interventions: Other: core muscle activation using physical fitness

INTERVENTIONS:
Other: core muscle activation using physical fitness — 2 instructors, they had physical therapy (PT) certificate, take an exam for subject's muscle strength of each muscle. After that time, subjects take a rest for 10 minutes. Researchers educate to subjects for high quality CPR including 5 to 6cm compression depth, 100 to 120 beat per minute (bpm) rate, complete chest recoil. Subjects perform chest compression to manikin with skill reporting system during 4min under guidance of 110 bpm metronome sound (first chest compression). After 1st chest compression, subjects take a rest during an hour and carry out PT. PT consist of 30 second plank for 3 sets, 12 times bridge for 3 sets and 20 times leg extension for 3 sets. Subjects take a rest during 30 seconds between sets, 1 minute every 3 sets.
  After PT completion, subjects take a rest during 10 minutes, and then perform 2nd chest compression in the same way of 1st chest compression. Researchers record subject's chest compression depth and rate in 1st and 2nd chest compression.
  Arms: after core muscle activation using physical fitness

SUMMARY:
Chest compression, a key component of cardiopulmonary resuscitation (CPR), has a major role for survival of cardiac arrest patients. According to 2015 American heart association (AHA) guideline, rescuers provide high quality CPR to adult cardiac arrest patients including 5 to 6 cm depth and 100 to 120 beat per minute rate chest compression.

However, in CPR situation, chest compression depth and rate vary according to provider's muscle strength. In other words, the individual difference of the degree of physical activity will make the different result for CPR. So, the investigators hypothesize that the core muscles activation using physical fitness improves the quality of chest compression and the quality of CPR, eventually.

ELIGIBILITY:
Inclusion Criteria:

* medical school students and interns had experienced in cardiopulmonary resuscitation (CPR) education

Exclusion Criteria:

* patients with musculoskeletal disease
* patients with cardiovascular disease
* patients with lung disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
mean chest compression depth | 1 Day

SECONDARY OUTCOMES:
the ratio of complete chest compression (5 to 6cm depth, complete chest recoil) to all chest compression | 1 Day

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, Seoul, South Korea